CLINICAL TRIAL: NCT01429272
Title: Minocycline and Aspirin in the Treatment of Bipolar Depression
Acronym: Minocycline
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Laureate Institute for Brain Research, Inc. (Other)
Collaborators: Stanley Medical Research Institute (Other); University of Oklahoma (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LIBR 2011-002
Record Dates: First submitted 2011-09-02; First posted 2011-09-07 (Estimated); Results first posted 2017-11-08 (Actual); Last update posted 2018-01-11 (Actual); Status verified 2017-12

CONDITIONS: Bipolar Disorder Depression
Keywords: Bipolar Disorder; Minocycline
MeSH Terms: conditions — Bipolar Disorder; cyclopia sequence | interventions — Minocycline; Aspirin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo & Placebo (Placebo Comparator): Placebo for minocycline & placebo for aspirin
  Interventions: Drug: placebo
- minocycline & aspirin (Active Comparator): Minocycline 100mg PO BID for 6 weeks & Aspirin 81 mg PO BID for 6 weeks
  Interventions: Drug: Minocycline; Drug: Aspirin

INTERVENTIONS:
Drug: Minocycline — 100 mg po bid for 6 weeks
  Arms: minocycline & aspirin
Drug: Aspirin — 81 mg po bid for 6 weeks
  Arms: minocycline & aspirin
Drug: placebo — placebo for minocycline and/or aspirin
  Arms: Placebo & Placebo

SUMMARY:
The purpose of this study is to determine whether minocycline and aspirin are effective in the treatment of depression in individuals with bipolar disorder.

DETAILED DESCRIPTION:
Abstract:

New medication classes are needed to improve treatment effectiveness in the depressed phase of bipolar disorder (BD). Extant evidence suggests that BD is not only characterized by reduced monoaminergic signaling, but also by neural changes such as dendritic remodeling, demyelination, and glial and neuronal cell loss. These changes have been hypothesized to result from chronic inflammation, based partly on convergent evidence that proinflammatory cytokines are elevated in depressed patients with BD. The principal aims of the proposed research is to evaluate the antidepressant efficacy in bipolar depression of minocycline, a drug with neuroprotective and immune-modulating properties, and of aspirin, at doses expected to selectively inhibit cyclooxygenase 1 (COX-1), within the context of a randomized, double-blind, placebo-controlled, parallel-group clinical trial following a 2 x 2 design.

Specific Aims Specific Aim 1: To evaluate the efficacy of augmentation therapy with minocycline and/or aspirin for bipolar depression.

The investigators will test the hypothesis that compared with placebo, participants receiving minocycline and/ or aspirin will show a greater treatment response rate (defined as a >50% increase on the MADRS for the final two consecutive visits).

Specific Aim 2: To investigate the relationship between the response to minocycline, aspirin and markers of inflammation (serum concentrations of IL-6 and CRP).

The investigators will test the hypotheses that: a) minocycline treatment will reduce inflammation to a greater extent than placebo; b) during minocycline treatment the change in inflammatory cytokine expression will correlate with the change in depression ratings; c) the baseline elevation of inflammatory markers will predict greater antidepressant response to minocycline.

ELIGIBILITY:
Inclusion Criteria:

One hundred and twenty male or female outpatients between 18 and 65 years of age, who meet DSM-IV-TR criteria for BD (type I or II or NOS) and for a current major depressive episode will be recruited. The depressive syndrome must have been present for at least 4 weeks and the minimum threshold for depression severity will be set at a Quick Inventory of Depressive Symptomatology (QID-C16) score >10. Subjects will provide written informed consent as approved by the Western Institutional Review Board.

Exclusion Criteria:

(a) Illness onset after 40 years of age; (b) serious risk of suicide; (c) current delusions or hallucinations sufficient to interfere with the capacity to provide informed consent; (d) current manic symptoms of sufficient severity to pose a substantial risk of the development of a manic episode; (e) current treatment with more than four psychotropic medications; (f) medical illness including hepatic impairment, renal dysfunction, bleeding diatheses, cerebrovascular disease, hypertension or diabetes mellitus that is inadequately controlled by diet and/or medication, or known active peptic ulcer disease; (g) abuse of drugs or alcohol within the preceding 6 months, or substance dependence within the last year; (h) daily alcoholic beverage consumption equivalent to >3 oz. of alcohol; (i) known allergies or hypersensitivities to tetracycline antibiotics, aspirin or other NSAIDs; (j) current use of drugs that could increase the risks associated with aspirin or minocycline administration, (k) chronic infection, (l) use of antibiotics, (m) pregnant or nursing women, (n) asthma which in the opinion of the investigator would increase the likelihood of an asthmatic attack, and (o) regular use of steroidal or non-steroidal anti-inflammatory medications (occasional use of NSAIDS was allowed).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2011-09; Primary Completion 2015-08 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sheldon Preskorn, MD, Principal Investigator — Laureate Institute for Brain Research, Inc.
Locations (3):
- United States (3):
  - University of Kansas Medical Center Research Institute, Wichita, Kansas
  - University of Oklahoma Department of Psychiatry, Tulsa, Oklahoma
  - Laureate Institute for Brain Research, Tulsa, Oklahoma

REFERENCES:
- [Derived] Savitz J, Preskorn S, Teague TK, Drevets D, Yates W, Drevets W. Minocycline and aspirin in the treatment of bipolar depression: a protocol for a proof-of-concept, randomised, double-blind, placebo-controlled, 2x2 clinical trial. BMJ Open. 2012 Feb 22;2(1):e000643. doi: 10.1136/bmjopen-2011-000643. Print 2012. PMID 22357572
- See also: Related Info — http://www.laureateinstitute.org/

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo + Minocycline: placebo aspirin + active minocycline
- Placebo + Aspirin: placebo minocycline + active aspirin
Period: Overall Study
Arm/Group | Placebo & Placebo | Minocycline & Aspirin | Placebo + Minocycline | Placebo + Aspirin
Started | 30 | 31 | 19 | 19
Completed | 24 | 22 | 15 | 14
Not Completed | 6 | 9 | 4 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo & Placebo | Minocycline & Aspirin | Placebo + Minocycline | Placebo + Aspirin | Total
Number analyzed (Participants) | 30 | 31 | 19 | 19 | 99
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 30 | 31 | 19 | 19 | 99
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 40.8 (10.4) | 40.8 (9.7) | 44.8 (8.7) | 40.6 (10.2) | 41.5 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 26 | 13 | 13 | 74
  Male | 8 | 5 | 6 | 6 | 25
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 30 | 31 | 19 | 19 | 99
Montgomery-Asberg Depression Rating Score [Mean (Standard Deviation); unit: units on a scale] — Range of scores (total) = 0-60. Higher scores indicate more depressive symptoms.
  units on a scale | 29.2 (6.2) | 28.0 (5.7) | 27.2 (5.2) | 25.9 (6.5) | 27.8 (5.9)
Measure of Inflammation using the C-Reactive Protein (CRP) measurement [Mean (Standard Deviation); unit: mg/L] — Measure of inflammation
  mg/L | 4.4 (5.3) | 8.2 (12.9) | 4.3 (5.5) | 4.5 (4.9) | 5.6 (8.5)
Interleukin 6 (IL-6) [Mean (Standard Deviation); unit: pg/ML] — Pro-inflammatory cytokine.
  pg/ML | 0.9 (0.5) | 1.0 (0.7) | 0.9 (0.5) | 1.1 (0.7) | 1.0 (0.6)

OUTCOME MEASURES:

1. Primary Outcome: Treatment Response
Description: Response to treatment defined as a >50% decrease in Montgomery-Asberg Depression Rating Scale scores for the final two consecutive visits.
Time Frame: Six weeks
Population: Note numbers do not match the participants flow because participants who did not return for at least one post treatment visit could not be included in the analysis.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo & Placebo | Minocycline & Aspirin | Placebo + Minocycline | Placebo + Aspirin
Number analyzed (Participants) | 28 | 30 | 18 | 19
Percentage of Participants | 21 | 44 | 25 | 50

2. Secondary Outcome: Remission Rate
Description: Remission defined as a score of <11 on Montgomery-Asberg Depression Rating Scale scores for the final two consecutive visits.
Time Frame: Six weeks
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Placebo & Placebo | Minocycline & Aspirin | Placebo + Minocycline | Placebo + Aspirin
Number analyzed (Participants) | 28 | 30 | 18 | 19
percentage of participants | 14 | 26 | 6 | 28

ADVERSE EVENTS:
Time Frame: Three years
Arm/Group | Placebo & Placebo | Minocycline & Aspirin | Placebo + Minocycline | Placebo + Aspirin
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/31 | 0/19 | 0/19
Other Adverse Events (participants affected / at risk) | 0/30 | 0/31 | 0/19 | 0/19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No